CLINICAL TRIAL: NCT05499000
Title: The Effect of Emotional Freedom Technique on Premenstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Sinem GUVEN Santur, Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Faculty of Health Science
Record Dates: First submitted 2022-08-07; First posted 2022-08-12 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Premenstrual Syndrome; Emotional Problem
Keywords: Emotional Freedom Technique; Premenstruel Sendrom; Midwifery
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Emotional freedom technique will be applied online with the researcher in 2 sessions, 3 days apart.
  KBF, SUE, PMSS pre-tests will be applied before the intervention, SUE will be applied before and after each session, At the end of the second session, post-test data will be obtained with SUE, PMSS.
  Interventions: Behavioral: Emotional freedom technique
- Control group (No Intervention): KBF, SUE and PMSS pre-tests will be applied to the participants, SUE, PMSS and post-test data will be obtained simultaneously with the experimental group.

INTERVENTIONS:
Behavioral: Emotional freedom technique — Emotional freedom technique will be applied online with the researcher in 2 sessions, 3 days apart.
  KBF, SUE, PMSS tests will be applied before the intervention, SUE will be applied before and after each session, At the end of the 2nd session, post-test data will be taken with SUE, PMSS.
  Arms: Experimental group

SUMMARY:
Objective: This study was conducted to evaluate the Effect of Emotional Freedom Technique on Premenstrual Syndrome.

Methodology: The research will be conducted as a randomized controlled trial. The research will be carried out with students studying at the Department of Midwifery, Faculty of Health Sciences, İnönü University, between September and October 2022. The sample size of the study was calculated as 102 people with an effect size of 0.80 and a power of 0.95. Premenstrual syndrome scale will be applied to all students participating in the research first and those who score 110 and above will be listed. Experimental and control groups will be determined by randomization. Personal information form, subjective experience unit scale and premenstrual syndrome scale will be used to collect data.

SPSS 22.0 package program will be used in the evaluation of the data. The independent variable of the research is the emotional liberation technique. The dependent variable of the study is the mean scores of the participants from the subjective experience unit scale and premenstrual syndrome scale.

DETAILED DESCRIPTION:
Menstruation is an important process accompanied by physiological and psychological fluctuations covering a long part of a woman's life. Premenstrual syndrome (PMS) is characterized by cyclical repetition of physical, psychological and behavioral symptoms that start one week before menstruation, gradually increasing in severity, and end with menstruation [1-3]. Presence of at least one of six affective symptoms (anger outburst, depression, anxiety, confusion, irritability, and social withdrawal) and one of four somatic symptoms (abdominal swelling, headache, breast tenderness, and swelling in the extremities) according to the American Association of Obstetricians and Gynecologists (ACOG). It states that if the symptoms disappear 4 days after the onset of the disease, and if it recurs cyclically, it meets the diagnostic criteria of PMS [4]. In studies conducted on PMS in various societies, its prevalence was determined to be in the range of 10-98% [5-8]. Although the etiology is not known exactly, the most common view is in the direction of serotonergic dysregulation. It is thought that the level of serotonin negatively affects the severity and intensity of PMS symptoms, and also triggers or exacerbates symptoms such as anxiety, appetite change and restlessness with the decrease in beta endorphin levels [9,10]. According to the severity level in PMS treatment; lifestyle changes (regular exercise, stress avoidance, regular sleep, etc.), combined oral contraceptives, serotonin selective inhibitors and cognitive behavioral therapies can be used [3, 11]. ACOG recommends using non-pharmacological treatments rather than pharmacological treatments for mild symptoms with psychological predominance [4].

Although it has a history of thousands of years in eastern cultures, it argues that the methods of energy psychology that we have encountered in the last 40 years in western societies and that psychological problems are related to disturbances in the energy fields of the body. According to energy psychology, people are physiological, emotional, mental and behavioral whole and in harmony. When the harmony is disturbed, psychological symptoms occur, and treatment is aimed by regulating the energy frequency by taking initiatives for this [12, 13]. In this context, Emotional Freedom Technique (EFT) is a psychophysiological method that provides easy and fast results to manage the normal energy flow on the energy body of the person [14, 15]. The main purpose of EFT is; It is to transform the negative energy frequency of the person into a positive one by clearing the negative emotions and thoughts that the person has subconsciously created or carried from the past by himself or environmental influences [14]. In the 1980s, thought field therapy, which was applied with strokes/touches to human meridian points with a complex algorithmic order, was simplified by Craig and started to apply with a single algorithmic order, thus EFT emerged [16, 17]. EFT is applied with strokes/touches as a somatic stimulus applied to meridian points, which includes stimulating the subconscious as in cognitive behavioral therapies, accepting a negative situation or emotion as in exposure therapy. It is frequently used in the treatment of psychological symptoms in current studies because it is easy to apply in opening the blockages in the energy body or converting the negative frequency to positive and has a quick result [18]. There are studies showing that EFT has positive effects on variables such as anxiety [14], phobias [15], posttraumatic stress disorder [16] and depression [17]. In the field of women's health, the effects of EFT studies on psychological development and cortisol levels in pregnant women with prenatal loss [18], fear of childbirth [19], dysmenorrhea [20] and postpartum depression [21] The results are extremely positive. In this context, it is thought that the research will contribute to the literature due to the insufficiency of studies examining the effect of EFT application on premenstrual syndrome.

ELIGIBILITY:
Inclusion Criteria:

* To be between 18-25,
* Single,
* Not to use anything pharmacological or non-pharmacological during the research,
* Not having a diagnosed psychiatric disease such as epilepsy.

Exclusion Criteria:

* Willingness to leave during research.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Subjective Units of Experience- (SUE) | Each participant will be evaluated for 1 week.
  The negative 10 feel the greatest pain, disappointment, fear, stress, sadness, or discomfort imaginable.
  When it reaches Positive 10, the client feels very different and wonderful. The meanings of the ratings in this range change gradually. The scale has no cutoff score. It is interpreted according to the mean of the scores and its relevance to other variables.

SECONDARY OUTCOMES:
Descriptive Data- (KBF) | It will be obtained in 1 week at the beginning of the research.
  The personal information form prepared by the researcher in line with the literature consists of socio-demographic (age, education and employment status, income status, family type and place of residence), obstetric (age of menarche, menstrual cycle duration), psycho-social and medical history questions.
Premenstrual Syndrome Scale- (PMSS) | It will take an average of 1 month to obtain the data. Measured PMSS scale data will be reported within 2 weeks at the end of the study.
  The reliability and validity study of the Premenstrual Syndrome Scale was performed by Gençdoğan (2006). The scale used to determine premenstrual symptoms and their severity is a 5-point Likert type and consists of 44 items. The scale has nine sub-dimensions: depressive affect, anxiety, irritability, fatigue, depressive thoughts, pain, changes in appetite and bloating. The lowest score that can be obtained from these nine sub-dimensions is 44, and the highest score is 220. A high score indicates that the intensity of premenstrual symptoms is high. The Cronbach alpha coefficient of the scale was found to be 0.75 (Gencdogan, 2006).

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha OZSAHİN, PhD, Study Director — https://www.inonu.edu.tr/akademik/zeliha.ozsahin; Yeşim AKSOY DERYA, PhD, Study Chair — https://www.inonu.edu.tr/akademik/yesim.aksoy; Çiğdem KARAKAYALI AY, PhD, Study Chair — https://saglikbilimleri.ozal.edu.tr/?page_id=7732
Locations (1):
- Inonu University Faculty of Health Sciences, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will be obtained by Personal Information Form, Subjective Experience Units (SUE), Premenstrual Syndrome Scale (PMSS).